CLINICAL TRIAL: NCT03330301
Title: D-tecting Disease - From Exposure to Vitamin D During Critical Periods of Life
Acronym: D-tect
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Council for Strategic Research (Other)
Responsible Party: Principal Investigator, Berit Lilienthal Heitmann, Professor, Bispebjerg Hospital
Other Study IDs: 0603-00453B
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Vitamin D Deficiency; Obesity; Diabetes Mellitus; Pre-Eclampsia; Arthritis; Asthma; Bone Fracture; Tooth Diseases; Birth Weight; Birth Disorder; Pregnancy Complications; Mental Disorder; Cancer; Congenital Disorders
MeSH Terms: conditions — Vitamin D Deficiency; Obesity; Diabetes Mellitus; Pre-Eclampsia; Arthritis; Asthma; Fractures, Bone; Tooth Diseases; Birth Weight; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Pregnancy Complications; Mental Disorders; Neoplasms | interventions — Cari-D-Tect

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 33 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: 1. Individuals born between June1983 and May1985 were exposed to the mandatory vitamin D margarine fortification during fetal life.
  2. Cases: individuals defined as having one of the aforementioned diseases of interest from the registers
  Interventions: Other: D-tect
- Non-exposed: 1. Individuals born between September1986 and August 1988 were not exposed to the mandatory vitamin D margarine fortification during fetal life.
  2. Controls: cohort of matched disease-free individuals
  Interventions: Other: D-tect

INTERVENTIONS:
Other: D-tect — 1. This study is based on a unique Danish social experiment that took place during a well-defined period between 1937 and December 1985, when it was mandatory to fortify all margarine with vitamin D (1.25 μg/100 g). This well-defined vitamin D fortification period makes it possible to investigate the impact of fetal exposure to extra vitamin D from food fortification on the risk of developing diseases later on. This study is possible due not only to the well-defined adjacent time window but also to the complete registration of every citizen via a civil registration number. This number can be linked, on an individual level, to Danish birth, patient and medical registries; social and ethnic registries; and clinical and other large databases
  2. Case-cohort study: vitamin D measurements from dried blood spots and the risk of diseases later on

SUMMARY:
Vitamin D deficiency is common among otherwise healthy pregnant women and may have consequences for them as well as the early development and long-term health of their children. However, the importance of maternal vitamin D status has not been widely studied.

The present study is divided into a societal experiment (1) and a case-cohort study (2):

1. The present study includes an in-depth examination of the influence of exposure to vitamin D early in life and during critical periods of growth for development of type 1 diabetes (T1D), type 2 diabetes, gestational diabetes, pre-eclampsia, obesity, asthma, arthritis, cancer, mental and cognitive disorders, congenital disorders, dental caries and bone fractures during child- and adulthood. The study is based on the fact that mandatory fortification of margarine with vitamin D, which initiated in 1937, was terminated in 1985.

   Apart from determining the influences of exposure prior to conception and during pre- and postnatal life, the investigators examined the importance of vitamin D exposure during specific seasons and trimesters, by comparing disease incidence among individuals born before and after the fortification.
2. Additionally, a validated method was used to determine neonatal vitamin D status using stored dried blood spots (DBS) from individuals who develop the aforementioned disease entities as adults and their time and gender-matched controls.

Unparalleled, the study will help determine the effects of vitamin D exposure during critical periods in life. There are a sufficient number of individuals to verify any effects during different gestation phases and seasons of the year. The results, which will change our current understanding of the significance of vitamin D, will enable new research in related fields, including interventional research designed to assess supplementation needs for different subgroups of pregnant women. Also, other health outcomes can subsequently be studied to generate multiple new interdisciplinary health research opportunities involving vitamin D.

ELIGIBILITY:
Inclusion Criteria:

1. Born in Denmark around the fortification period
2. Sufficient amount of blood from the DBS

Exclusion Criteria:

1.Born outside Denmark

1. Born outside the fortification period
2. Insufficient amount of blood from the DBS or DBS not found

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Entire Danish population born between June1983-May1985 and September 1986-August 1988.
  For the part of the study using vitamin D measurements from DBS:
  The Danish Civil registration system was used to identify all live-born children during 1981-2002 (n = 1,360,466), and a random subcohort thereof was sampled for 25(OH)D analyses to be used across the D-tect studies (n = 3585)
Sampling Method: Probability Sample
Enrollment: 222776 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Obesity | 2012-2025
  Register based
Type 1 diabetes | 2012-2016
  Register based
Pre-eclampsia | 2012-2025
  Register based
Bone facture | 2012-2025
  Register based

SECONDARY OUTCOMES:
Type 2 diabetes | 2014-2025
  Register based
Gestational diabetes | 2014-2025
  Register based
Asthma | 2015-2025
  Register based
Arthritis | 2018-2025
  Register based
Birth weight | 2014-2019
  Register based
Mental diseases | 2012-2025
  Register based

OTHER OUTCOMES:
Cancers | 2018-2025
  Register based
Mental disorders | 2018-2025
  Register based
Dental caries | 2018-2025
  Register based
Congenital disorders | 2018-2025
  Register based

CONTACTS AND LOCATIONS:
Locations (1):
- Parker Institute, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keller A, Stougard M, Frederiksen P, Thorsteinsdottir F, Vaag A, Damm P, Jacobsen R, L Heitmann B. In utero exposure to extra vitamin D from food fortification and the risk of subsequent development of gestational diabetes: the D-tect study. Nutr J. 2018 Nov 2;17(1):100. doi: 10.1186/s12937-018-0403-5. PMID 30388966
- See also: Study website — http://www.d-tectingdisease.dk/